CLINICAL TRIAL: NCT05634083
Title: Does Indoxyl Sulfate Have a Role in Uremic Pruritus? A Laboratory and Interventional Study.
Brief Title: Does Indoxyl Sulfate Have a Role in Uremic Pruritus?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Essam Mohamed El-sayed Akl, Assistant Professor of Dermatology and Andrology, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC 22-10-2022
Record Dates: First submitted 2022-11-18; First posted 2022-12-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: Patients will take activated charcoal for two months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uremic Pateints group (Experimental): Patients with end-stage renal failure with itching
  Interventions: Dietary Supplement: Uremic pateints with itching

INTERVENTIONS:
Dietary Supplement: Uremic pateints with itching — Activated charcoal

SUMMARY:
Itching is a widespread and disturbing complain from patients with chronic kidney disease (CKD); epidemiologic data have suggested that approximately 40% of patients with end-stage renal disease experience moderate to severe itching. The pathogenesis of renal pruritus is multifactorial. Triggering factors may include uremia-related abnormalities, accumulation of uremic toxins, systemic inflammation and cutaneous xerosis. Indoxyl sulfate (IS) is a protein-bound uremic toxin resulting from the metabolism of dietary tryptophan accumulating in patients with end-stage renal disease.

DETAILED DESCRIPTION:
Patients with end-stage renal disease undergoing hemodialysis complaining of itching not related to other cause than renal failure will take activated charcoal with foods and serum level of indoxyl sulphate will be studied

ELIGIBILITY:
Inclusion Criteria:

Patients with end-stage renal failure with itching undergoing regular hemodialysis

Exclusion Criteria:

Patients with other causes of itching as psoriasis, atopic dermatitis, scabies, and lichen planus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Severity of itching | Two months
  Change of severity of itching by The Visual Analogue Scale score

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Benha University, Al Qalyūbīyah, Benha
  - Benha University Hospitals, Banhā

IPD SHARING:
Plan to Share IPD: No